CLINICAL TRIAL: NCT04414696
Title: Preventing Postpartum Depression: Exercise as Medicine
Brief Title: Postpartum Wellness
Acronym: POW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1548855
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Depression
Keywords: Exercise; Postpartum Depression; Physical activity; eHealth intervention
MeSH Terms: conditions — Depression, Postpartum; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Investigators and programmers/analysts will be blinded to the intervention assignment. The participants, project manager and research assistant will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be asked to use a web-based (eHealth) exercise intervention for 3 months. This eHealth exercise intervention includes over 90, 10-minute exercise videos with options for exercise type, time, and intensity, customized to the weight of the infant. Users can either select up to three 10-minute videos to create a 10 to 30-minute workout or choose a 'Ready Made' workout that is either 10, 20, or 30-minutes long.
  Interventions: Behavioral: Exercise intervention
- Usual Care (No Intervention): Participants in the usual care condition will follow their usual standard care as suggested by their provider. Participants will complete the same assessments and incentives as the active intervention but will not receive the eHealth exercise intervention.

INTERVENTIONS:
Behavioral: Exercise intervention — eHealth exercise intervention for postpartum women at increased risk of depression
  Arms: Intervention

SUMMARY:
The purpose of this study is to test whether a web-based (eHealth) exercise intervention for new moms at increased risk for postpartum depression increases physical activity and decreases postpartum depression symptoms.

DETAILED DESCRIPTION:
Postpartum depression is a debilitating and costly condition that is associated with significant health consequences for mothers and children. Counseling for prevention of postpartum depression is currently recommended in women at high risk of postpartum depression; however, there is a shortage of mental health care providers. There is a need for effective interventions to prevent postpartum depression that can be easily integrated into health care systems, yet do not involve intense health care system resources. eHealth interventions are promising in this regard.

Strong evidence suggests physical activity can reduce depression risk. This study will assess the effectiveness of an eHealth exercise intervention tailored to postpartum mothers for increasing physical activity levels and improving depressive symptoms in women at increased risk of postpartum depression. This intervention addresses several identified barriers to physical activity in postpartum women. The study will randomize 200 women to receive an eHealth exercise intervention for postpartum women or usual postpartum care. Device-based physical activity and depressive symptoms will be measured at 3 and 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* KPNC member between 2 and 6 months postpartum
* Current PHQ-8 score between 10-20 and no current depression diagnosis
* Delivered baby in KPNC
* English-speaking
* Own a smartphone, computer, or TV with internet access
* Free of a heart condition and a physician recommending medically supervised physical activity
* Body Mass Index (BMI) between 18.5 and 40 (kg/m2)
* A baby weighing between 11-22 lbs

Exclusion Criteria:

* Engaged in regular, moderate or vigorous physical activity >90 minutes or more per week
* Pregnant or planning to become pregnant in the ensuing three months
* A baby with chronic illness/disorder(s) that prevent participant from holding or lifting him/her
* Chest pain during physical activity, or has had chest pain within the prior month
* Taking medication for hypertension or a heart condition
* Tendency to fall due to syncope or dizziness
* Orthopedic problems that might be aggravated by physical activity
* Has exercise-induced asthma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsay Avalos, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramsey M, Oberman N, Quesenberry CP Jr, Kurtovich E, Gomez Chavez L, Chess A, Brown SD, Albright CL, Bhalala M, Badon SE, Avalos LA. A Tailored Postpartum eHealth Physical Activity Intervention for Individuals at High Risk of Postpartum Depression-the POstpartum Wellness Study (POW): Protocol and Data Overview for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 29;13:e56882. doi: 10.2196/56882. PMID 39470705

RESULTS

PARTICIPANT FLOW:
Period: 3-month Follow up
Arm/Group | Intervention | Usual Care
Started | 50 | 49
Completed | 27 | 26
Not Completed | 23 | 23
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 22 | 23
Period: 6-month Follow up
Arm/Group | Intervention | Usual Care
Started | 27 | 26
Completed | 21 | 22
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (5.1) | 32.7 (4.5) | 32.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 6 | 4 | 10
  Hispanic | 10 | 12 | 22
  Non-Hispanic Black | 3 | 3 | 6
  Non-Hispanic White | 19 | 18 | 37
  Other | 12 | 12 | 24
Months postpartum [Mean (Standard Deviation); unit: months] | 4.1 (1.2) | 4 (1) | 4.1 (1.1)
Number of children at home [Count of Participants; unit: Participants]
  2+ | 30 | 28 | 58
  1 | 20 | 21 | 41
Depressive symptons [Mean (Standard Deviation); unit: score on a scale] — Continuous measure of depressive symptoms as assessed using the Patient Health Questionnaire (PHQ-8).
  PHQ-8 scores range from 0-24. A score of 1-4 suggests minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression and 20-24 severe depression.
  score on a scale | 12.6 (2.2) | 12.6 (2.2) | 12.6 (2.2)
Physical activity level prior to pregnancy [Count of Participants; unit: Participants] — Measured using the Stanford Leisure-Time Activity Categorical Item (L-Cat) modified to reflect the year before pregnancy
  Participants
    Below recommendations | 29 | 31 | 60
    At or above recommendations | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms
Description: Continuous measure of depressive symptoms as assessed using the Patient Health Questionnaire (PHQ-8).
  PHQ-8 scores range from 0-24. A score of 1-4 suggests minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression and 20-24 severe depression.
Time Frame: 3 months
Population: After multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale | 10.1 (5.4) | 11 (5.8)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.3 to 1.5] — Multivariable linear regression

2. Primary Outcome: Device-Measured Physical Activity
Description: Actigraph-measured minutes of moderate/vigorous physical activity
Time Frame: 3 months
Population: After multiple imputation
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
minutes per day | 53.2 (39.9) | 58 (44.8)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-23.5 to 14.5] — Multivariable linear regression

3. Secondary Outcome: Self-reported Physical Activity
Description: Self-reported moderate/vigorous physical activity
Time Frame: 3 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: MET-hours per week
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
MET-hours per week | 15.8 (15.7) | 12.7 (14.7)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-1.9 to 9.5]

4. Secondary Outcome: Device-measured Physical Activity
Description: Actigraph-measured minutes of moderate/vigorous physical
Time Frame: 6 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
minutes per day | 63.2 (49.1) | 62.3 (53.8)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-18.9 to 21.5] — Multivariable linear regression

5. Secondary Outcome: Depressive Symptoms
Description: Continuous measure of depressive symptoms as assessed in the Patient Health Questionnaire (PHQ-8).
  PHQ-8 scores range from 0-24. A score of 1-4 suggests minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression and 20-24 severe depression.
Time Frame: 6 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale | 7.9 (4.9) | 9.1 (5.4)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.7 to 1.1] — Multivariable linear regression

6. Secondary Outcome: Self-reported Physical Activity
Description: Self-reported moderate/vigorous physical activity
Time Frame: 6 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: MET-hours per week
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
MET-hours per week | 13.7 (13.8) | 16.3 (16.6)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.7 to 4.2] — Multivariable linear regression

7. Other Pre Specified Outcome: Sleep
Description: Sleep quality measured using the Pittsburgh Sleep Quality Index (PSQI).
  The Pittsburgh Sleep Quality Index (PSQI) asks about sleep quality during the past month, including questions on sleep duration, sleep disturbance, and use of sleep-inducing medications. A global score, ranging from 0 to 21, is calculated using seven components of sleep. Higher scores indicate poorer sleep quality.
Time Frame: 3 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale | 9.6 (4) | 10.1 (4.2)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.2 to 2.1] — Multivariable linear regression

8. Other Pre Specified Outcome: Mother-infant Bonding
Description: The Mother Infant Bonding Scale will be used to assess mother-infant bonding.
  Mother Infant Bonding Scale scores range from 0-24. Higher scores indicate worse mother-infant bonding.
Time Frame: 3 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale | 1.7 (2.9) | 1.8 (3)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1.1] — Multivariable linear regression

9. Other Pre Specified Outcome: Anxiety
Description: The General Anxiety Disorder Scale (GAD-7) will be used to assess anxiety.
  GAD-7 scores range from 0-21. A score of 1-4 suggests minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.
Time Frame: 3 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale | 9.2 (5.4) | 10 (5.7)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.4 to 1.2] — Multivariable linear regression

10. Other Pre Specified Outcome: Stress
Description: Perceived stress will be measured using the Perceived Stress Scale (PSS-10).
  PSS-10 scores range from 0-40 with higher scores indicating higher perceived stress. A score of 0-13 suggests low stress, 14-26 moderate stress, and 27-40 high perceived stress.
Time Frame: 3 months
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale | 21 (6.7) | 23.2 (7.3)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.9 to 1.3] — Multivariable linear regression

11. Other Pre Specified Outcome: Infant Development
Description: Ages and Stages questionnaire for 12-month-old infants.
  The ASQ-3 screens for delays in infant and child development in five domains: communication, gross motor, fine motor, problem-solving, and personal adaptive skills. Scores for each of the five domains range from 0-60 with higher scores indicating typical development.
Time Frame: At 12 months old
Population: Intent to treat analysis with multiple imputation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
score on a scale
  Communication | 44.6 (13.9) | 42.1 (14.7)
  Gross motor function | 47.6 (15.1) | 47.5 (14.5)
  Fine motor function | 50 (9.4) | 48.5 (9.5)
  Problem-solving | 42 (12.9) | 41.1 (13.8)
  Personal-social skills | 40.1 (13.5) | 36.9 (14)

ADVERSE EVENTS:
Time Frame: 6 months of follow up
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04414696/Prot_SAP_000.pdf